CLINICAL TRIAL: NCT05507307
Title: The Effect of Mindfulness-Based Pregnancy Education Program on Stress, Birth Fear and Birth Self-Efficacy in Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sıdıka Özlem CENGİZHAN, Assistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117.17.06
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Mindfulness; Pregnancy; Stress; Childbirth; Midwife

STUDY DESIGN:
Intervention Model Description: Randomized
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR group (Experimental): mindfulness-based pregnancy education program group
  Interventions: Behavioral: mindfulness-based pregnancy education program.
- Control group (No Intervention): control group standard care group

INTERVENTIONS:
Behavioral: mindfulness-based pregnancy education program. — Pregnant education program based on mindfulness is planned as 2 sessions per week for 4 weeks, in total 8 sessions. Each session is planned to last 40-60 minutes on average. Sessions will continue as individu
  Arms: MBSR group

SUMMARY:
The research will be carried out to determine the effect of mindfulness-based pregnancy education program on stress, fear of childbirth and birth self-efficacy in pregnant women. The study was designed as a randomized controlled trial. The universe of the research will consist of pregnant women who applied to Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital Pregnancy training class. The sample of the research, on the other hand, was determined by power analysis, at least the number of individuals to be included in the sample of the research. Sample size when power analysis is done; Assuming that the method applied with 5% error level, bidirectional significance level, 95% confidence interval and 80% ability to represent the universe, would reduce the anxiety score averages (30.53±6.49) by 4 points, a total of 84 pregnant women (42 experimental, 42 control) were calculated. Introductory Information Form", "Prenatal Distress Scale (PBL)-Revised Version", "Birth Attitude Scale" and "Birth Self-Efficacy Scale short form" will be used.

It is predicted that the research will contribute to the literature in line with its originality and results.

DETAILED DESCRIPTION:
The research will be carried out to determine the effect of mindfulness-based pregnancy education program on stress, fear of childbirth and birth self-efficacy in pregnant women. The study was designed as a randomized controlled trial. The universe of the research will consist of pregnant women who applied to Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital Pregnancy training class. The sample of the research, on the other hand, was determined by power analysis, at least the number of individuals to be included in the sample of the research. Sample size when power analysis is done; Assuming that the method applied with 5% error level, bidirectional significance level, 95% confidence interval and 80% ability to represent the universe, would reduce the anxiety score averages (30.53±6.49) by 4 points, a total of 84 pregnant women (42 experimental, 42 control) were calculated. Introductory Information Form", "Prenatal Distress Scale (PBL)-Revised Version", "Birth Attitude Scale" and "Birth Self-Efficacy Scale short form" will be used.

Pregnant Information Form: It is a form consisting of 21 questions developed by the researchers in line with the literature in order to determine the socio-demographic, obstetric and health characteristics of women.

Prenatal Distress Scale (PBL)- Revised Version The "Prenatal Distress Scale" was developed by Yali and Lobel in 1999 to assess women's social relations, physical and emotional symptoms, and concerns about themselves and their baby during pregnancy (14). The first 12-item scale was developed by Lobel in 2008 and a 17-item Prenatal Distress - Revised version was created (15). The Turkish validity and reliability study was performed by Yüksel et al. in 2011 (16). In the internal consistency analysis of the scale (n=522), the Cronbach's alpha internal consistency coefficient was 0.85, and the item 36 total score correlation coefficients (r) ranged from 0.20 to 0.78 (p<0.001). The scale is in 3-point Likert type. The participants are asked to read the statement in the scale and choose the one that suits them from the sequential statements "Not at all" (0), "A little" (1) and "Too much" (2). The minimum score that can be obtained from the scale is "0" and the maximum score is "34", and as the score obtained from the scale increases, prenatal distress levels also increase. The scale has no breakpoints.

Birth Attitude Scale Birth attitude scale is a scale developed by Lowe to measure fear of birth. This scale is a four-point Likert scale consisting of 16 items, with a high score indicating high anxiety. 1= No worries; no fear, 2= Low anxiety; not enough to be called fear, 3= moderate anxiety; distressing but enough to affect feelings of well-being 4 = high anxiety; It is evaluated as very worrying and affecting the sense of well-being. The Cronbach alpha coefficient of the scale, which was performed by Dönmez et al. in 2012, was found to be 0.82.

Birth Self-Efficacy Scale Short form The Birth Self-Efficacy Scale, consisting of 28 items, has two sub-dimensions as result expectation and self-efficacy expectation, scored from 1 to 10, 1 = 'I'm NOT SURE' 10 = 'TOTALLY SURE'. The lowest score that can be obtained from the scale is 28, the lowest The high score is 280, and it is accepted that as the score increases, birth self-efficacy increases, and as the score decreases, it decreases. Its Turkish validity and reliability were evaluated in 2021 by Aydın et al. The Cronbach alpha coefficient of the scale was found to be 0.82.

Data Collection: The data will be interviewed and invited by the researchers to the pregnant women who applied to the pregnant training class at Gaziantep Cengiz Gökçek Gynecology and Childhood Hospital between July 2022 and December 2022. Pregnant women who accept to participate in the study and meet the criteria will be filled by the researchers by face-to-face interview method. As a pre-test, "Descriptive Information Form", "Prenatal Distress Scale (PBL) - Revised Version", "Birth attitude scale" and "birth self-efficacy scale - short form" will be applied to the pregnants in the experimental and control groups. After the conscious awareness-based pregnancy education program was applied to the experimental group, 2 sessions a week for 4 weeks (1 month), a total of 8 sessions, the "Prenatal Distress Scale (PBL) - Revised Version", "Birth Attitude Scale" was applied to the experimental group and simultaneously to the control group. and 'birth self-efficacy scale-short form' will be applied. They will receive the pregnant training given in the routine pregnant class.

It is predicted that the research will contribute to the literature in line with its originality and results.

ELIGIBILITY:
Inclusion Criteria:

* Not having any diagnosed psychiatric disease,

  * Able to read and write,
  * Using a smart phone,
  * with internet access
  * Having a headset accessory for phone calls,
  * Pregnant women who voluntarily agreed to participate in the study

Exclusion Criteria:

* Pregnant women with communication barriers and mental disabilities
* Pregnant women under the age of 18

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Prenatal Distress Scale (PBL)- Revised Version | Change in stress at 4 weeks
  The "Prenatal Distress Scale" was developed by Yali and Lobel in 1999 to assess women's social relations, physical and emotional symptoms, and concerns about themselves and their baby during pregnancy (14). The first 12-item scale was developed by Lobel in 2008 and a 17-item Prenatal Distress - Revised version was created (15). The Turkish validity and reliability study was performed by Yüksel et al. in 2011 (16). In the internal consistency analysis of the scale (n=522), Cronbach's alpha internal consistency coefficient was 0.85, and item 36 total score correlation coefficients (r) ranged from 0.20 to 0.78 (p<0.001). The scale is 3-point Likert type.

SECONDARY OUTCOMES:
Birth Attitude Scale | Change in Birth Attitude within 4 weeks
  The birth attitude scale is a scale developed by Lowe to measure the fear of birth. This scale is a four-point Likert scale consisting of 16 items, with a high score indicating high anxiety. 1= No worries; no fear, 2= Low anxiety; not enough to be called fear, 3= moderate anxiety; distressing but enough to affect feelings of well-being 4 = high anxiety; It is evaluated as very worrying and affecting the sense of well-being. The Cronbach alpha coefficient of the scale, which was performed by Dönmez et al. in 2012, was found to be 0.82.

OTHER OUTCOMES:
Birth Self-Efficacy Scale Short form | Change in Birth Self-Efficacy within 4 weeks
  The Birth Self-Efficacy Scale, consisting of 28 items, has two sub-dimensions as result expectation and self-efficacy expectation, scored from 1 to 10, 1 = 'I'm NOT SURE' 10 = 'TOTALLY SURE'. The lowest score that can be obtained from the scale is 28, the lowest The high score is 280, and it is accepted that as the score increases, birth self-efficacy increases, and as the score decreases, it decreases. Its Turkish validity and reliability were evaluated in 2021 by Aydın et al. The Cronbach alpha coefficient of the scale was found to be 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Sıdıka Özlem CENGİZHAN, Assistant Professor, Principal Investigator — Gaziantep Islamic Science and Technology University faculty of health sciences
Locations (1):
- Faculty of Health Science, Gaziantep, Şahinbey/ Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne J, Hauck Y, Fisher C, Bayes S, Schutze R. Effectiveness of a Mindfulness-Based Childbirth Education pilot study on maternal self-efficacy and fear of childbirth. J Midwifery Womens Health. 2014 Mar-Apr;59(2):192-7. doi: 10.1111/jmwh.12075. Epub 2013 Dec 10. PMID 24325752
- [Background] Zemestani M, Fazeli Nikoo Z. Effectiveness of mindfulness-based cognitive therapy for comorbid depression and anxiety in pregnancy: a randomized controlled trial. Arch Womens Ment Health. 2020 Apr;23(2):207-214. doi: 10.1007/s00737-019-00962-8. Epub 2019 Apr 13. PMID 30982086
- [Background] Fenwick J, Toohill J, Gamble J, Creedy DK, Buist A, Turkstra E, Sneddon A, Scuffham PA, Ryding EL. Effects of a midwife psycho-education intervention to reduce childbirth fear on women's birth outcomes and postpartum psychological wellbeing. BMC Pregnancy Childbirth. 2015 Oct 30;15:284. doi: 10.1186/s12884-015-0721-y. PMID 26518597